CLINICAL TRIAL: NCT01290315
Title: A Randomized, Controlled Study to Investigate the Safety and Oxidative Stress Potential of Intravenous Ferric Carboxymaltose (FCM) vs. IV Iron Sucrose or IV Iron Dextran in Treating Iron Deficiency Anemia in Women
Brief Title: Intravenous Ferric Carboxymaltose vs IV Iron Sucrose or IV Iron Dextran in Treating Iron Deficiency Anemia in Women
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: American Regent, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1VIT08022
Record Dates: First submitted 2010-11-10; First posted 2011-02-07 (Estimated); Results first posted 2018-02-08 (Actual); Last update posted 2018-02-08 (Actual); Status verified 2018-02

CONDITIONS: Iron Deficiency Anemia
MeSH Terms: conditions — Anemia, Iron-Deficiency | interventions — ferric carboxymaltose; Ferric Oxide, Saccharated; Iron-Dextran Complex

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ferric Carboxymaltose (FCM) (Experimental): Intravenous iron
  Interventions: Drug: Ferric Carboxymaltose (FCM)
- Iron Sucrose / Iron Dextran (Active Comparator): Intravenous iron
  Interventions: Drug: Iron Sucrose / Iron Dextran

INTERVENTIONS:
Drug: Ferric Carboxymaltose (FCM) — One 500 mg dose at 100 mg/minute (Cohort I) or 750 mg dose at 100 mg/minute (Cohort II)
  Other Names: Injectafer
  Arms: Ferric Carboxymaltose (FCM)
Drug: Iron Sucrose / Iron Dextran — One 500 mg dose of IV iron sucrose administered over 4 hours (Cohort I), or a 750 mg dose of IV iron dextran administered as a 25 mg test dose over 5 minutes followed by a 725 mg dose over 3 hours if no adverse reaction to test dose is observed after 60 minutes (Cohort II)
  Other Names: Venofer, Dexferrum
  Arms: Iron Sucrose / Iron Dextran

SUMMARY:
The purpose of this study is to compare safety and the oxidative stress potential of two doses of an investigational IV iron, ferric carboxymaltose (FCM), compared to an equal single dose of IV iron sucrose or IV iron dextran in the treatment of Iron Deficiency Anemia (IDA) in female subjects.

DETAILED DESCRIPTION:
This was a Phase 2a, open-label, multicenter, randomized study that compared the safety and oxidative stress potential of FCM vs. IV iron sucrose or IV iron dextran in female subjects with IDA. Subjects with a diagnosis of IDA who required iron supplementation met all inclusion and no exclusion criteria, and had given informed consent were randomized. The duration of the study for each subject was a maximum of 6 weeks.

Eligible subjects were randomized in a 1:1 ratio to FCM (Group A) or IV iron sucrose or IV iron dextran (Group B).

Group A subjects received a single undiluted dose of iron as FCM by a slow IV injection on Day 0. Cohort I received 500 mg and Cohort II received 750 mg. Group B subjects received a single dose of iron as IV iron sucrose or as IC iron dextran on Day 0. Cohort I receive 500 mg iron sucrose and Cohort II received 750 mg iron dextran. Iron dextran administration was preceded by a 25 mg test dose 1 hour prior to infusion.

All subjects had laboratory assessments at Baseline, 2 hours post-infusion, 24 hours post-infusion, Day 7 (drawn at the same time of day [within 4 hours] as the 24-hour visit), and Day 30 (drawn at the same time of day [within 4 hours] as the the 24-hour visit). On Days 7 and 30, the safety evalutation for all subjects included treatment-emergent adverse event reporting, concomitant medication review, physical examination including vital signs, and laboratory assessments. Any subject who withdrew from the study received a follow-up phone call 30 days after they received study drug.

ELIGIBILITY:
Inclusion Criteria:

* Female subjects 18-50 years of age and able to give informed consent.
* If post-partum, at least 10 days post delivery at Day 0.
* Screening Visit local laboratory Hgb < or = to 10 g/dL or < or = to 12 g/dL with symptoms (dizziness and/or fatigue).
* Screening Visit ferritin < or = to 100 ng/mL or < or = to 300 when TSAT is < or = to 30%.
* Documented unsatisfactory response or intolerance to oral iron.

Exclusion Criteria:

* Previous participation in a ferric carboxymaltose (FCM) clinical trial.
* Known hypersensitivity reaction to any component of ferric carboxymaltose, Venofer, or Dexferrum.
* History of drug allergy or any history of rheumatoid arthritis or other autoimmune diseases.
* Current anemia not attributed to iron deficiency.
* During the 10 day period prior to screening has been treated with antibiotics.
* During the 30 day period prior to screening or during the study period has or will be treated with erythropoiesis stimulating agents.
* Active malignancy within 5 years. Basal or squamous cell skin cancer is not exclusionary.
* During the 30 day period prior to screening or during the study period has or will require a surgical procedure that necessitates general anesthesia.
* Current (acute or chronic) infection other than viral upper respiratory tract infection.
* AST or ALT at screening greater than 1.5 times the upper limit of normal.
* Known positive hepatitis B with evidence of active hepatitis.
* Known positive HIV-1/HIV-2 antibodies (anti-HIV).
* Patient has an active diagnosis of asthma and is currently using an anti- asthmatic therapy.
* Received an investigational drug within 30 days of screening.
* Alcohol or drug abuse within the past 6 months.
* Hemochromatosis or other iron storage disorders.
* Systolic blood pressure > or = to 180 or < 80 mmHg or diastolic blood pressure > or = to 100 or < 40 mmHg at screening or Day 0.
* Chronic kidney disease.
* Chronic inflammatory condition including but not limited to Lupus and Rheumatoid Arthritis.
* Pre-term delivery < 32 weeks.
* Emergent C-section delivery.
* Significant cardiovascular disease, including but not limited to myocardial infarction or unstable angina within 6 months prior to study inclusion or current history of NYHA Class III or IV congestive heart failure.
* Any other laboratory abnormality, medical condition or psychiatric disorder which in the opinion of the investigator puts the subject's disease management at risk or may result in the subject being unable to comply with study requirements.
* Night shift workers.
* Breastfeeding planned on or after Day 0.
* Pregnant or sexually-active female subjects who are of childbearing potential and who don't use an acceptable form of contraception.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 49 (Actual)
Dates: Start 2009-08 (Actual); Primary Completion 2013-03 (Actual); Study Completion 2013-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Linda M Mundy, MD, PhD, Study Director — American Regent, Inc.
Locations (1):
- Luitpold Pharmaceuticals, Inc., Norristown, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Hospitals and Medical Clinics. December 6, 2010 through October 13, 2012.
Pre-assignment Details: Discontinuation prior to dosing included lost to follow-up, subject request, and selection criteria/study compliance. A total of 19 subjects were excluded from the population of subjects evaluated for efficacy and safety-5 randomized to FCM 500mg, 2 randomized to FCM 750mg, 6 randomized to iron sucrose 500mg, and 6 randomized to iron dextran 750mg.
Groups:
- Ferric Carboxymaltose (FCM) Cohort I: Intravenous iron
  Ferric Carboxymaltose (FCM): One 500 mg dose at 100 mg/minute (Cohort I)
- Iron Sucrose Cohort I: Intravenous iron
  Iron Sucrose: One 500 mg dose of IV iron sucrose administered over 4 hours (Cohort I)
- Ferric Carboxymaltose (FCM) Cohort II: Intravenous iron
  Ferric Carboxymaltose (FCM): One 750 mg dose at 100 mg/minute (Cohort II)
- Iron Dextran Cohort II: Intravenous iron
  Iron Dextran: One 750 mg dose of IV iron dextran administered as a 25 mg test dose over 5 minutes followed by a 725 mg dose over 3 hours if no adverse reaction to test dose is observed after 60 minutes (Cohort II)
Period: Overall Study
Arm/Group | Ferric Carboxymaltose (FCM) Cohort I | Iron Sucrose Cohort I | Ferric Carboxymaltose (FCM) Cohort II | Iron Dextran Cohort II
Started | 14 | 12 | 10 | 13
Completed | 11 | 9 | 10 | 8
Not Completed | 3 | 3 | 0 | 5
Not completed — Adverse Event | 0 | 0 | 0 | 3
Not completed — Selection criteria/compliance | 2 | 1 | 0 | 2
Not completed — Lost to Follow-up | 0 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ferric Carboxymaltose (FCM) Cohort I | Iron Sucrose Cohort I | Ferric Carboxymaltose (FCM) Cohort II | Iron Dextran Cohort II | Total
Number analyzed (Participants) | 14 | 12 | 10 | 13 | 49
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 14 | 12 | 10 | 13 | 49
  >=65 years | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.1 (7.66) | 29.6 (9.93) | 39.2 (7.97) | 39.2 (9.21) | 34.8 (9.48)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 12 | 10 | 13 | 49
  Male | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 14 | 12 | 10 | 13 | 49

OUTCOME MEASURES:

1. Primary Outcome: Changes From Baseline in Markers of Oxidative Stress (Carbonyl and 8-isoprostane)
Time Frame: Change from Baseline to Day 30
Population: Only subjects with both a Baseline and at least one post-Baseline value are included.
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | Ferric Carboxymaltose (FCM) Cohort I | Iron Sucrose Cohort I | Ferric Carboxymaltose (FCM) Cohort II | Iron Dextran Cohort II
Number analyzed (Participants) | 12 | 9 | 10 | 10
mg
  Carbonyl | -11.90 (52.55) | -1.06 (38.722) | -12.37 (32.91) | -11.14 (48.57)
  8-isoprostane | 141.46 (892.16) | -369.50 (957.06) | 8.83 (81.20) | 32.28 (233.41)

2. Primary Outcome: Changes From Baseline in Markers of Oxidative Stress (Carbonyl and 8-isoprostane)
Time Frame: Change from baseline to 2 hours post end IV infusion
Population: Only subjects with both a baseline and at least one post baseline value are included.
Measure: Mean (Standard Deviation); unit: mg
Groups:
- Ferric Carboxymaltose (FCM) Cohort II: Intravenous iron
  Ferric Carboxymaltose (FCM): One 750mg dose at 100 mg/minute (Cohort II)
Arm/Group | Ferric Carboxymaltose (FCM) Cohort I | Iron Sucrose Cohort I | Ferric Carboxymaltose (FCM) Cohort II | Iron Dextran Cohort II
Number analyzed (Participants) | 12 | 10 | 10 | 11
mg
  Carbonyl: number analyzed (Participants) | 12 | 9 | 9 | 11
  Carbonyl | 2.07 (38.21) | 6.05 (24.69) | -8.66 (43.15) | -5.98 (23.71)
  8-isoprostane: number analyzed (Participants) | 12 | 9 | 9 | 11
  8-isoprostane | 151.59 (833.75) | -420.02 (803.52) | -2.64 (30.44) | -5.92 (216.66)

3. Primary Outcome: Changes From Baseline in Markers of Oxidative Stress (Carbonyl and 8-isoprostane)
Time Frame: Change from baseline to 24 hours post end IV infusion
Population: Only subjects with both a baseline and at least one post baseline value are included.
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | Ferric Carboxymaltose (FCM) Cohort I | Iron Sucrose Cohort I | Ferric Carboxymaltose (FCM) Cohort II | Iron Dextran Cohort II
Number analyzed (Participants) | 12 | 10 | 10 | 11
mg
  Carbonyl: number analyzed (Participants) | 11 | 10 | 9 | 11
  Carbonyl | 8.63 (23.24) | -6.92 (21.49) | 8.94 (87.05) | -11.57 (40.30)
  8-isoprostane: number analyzed (Participants) | 11 | 10 | 9 | 11
  8-isoprostane | 198.67 (864.29) | 119.26 (575.29) | -23.96 (60.01) | 38.02 (190.07)

4. Primary Outcome: Changes From Baseline in Markers of Oxidative Stress (Carbonyl and 8-isoprostane)
Time Frame: Change from baseline to Day 7 post end IV infusion
Population: Only subjects with both a baseline and at least one post baseline value are included.
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | Ferric Carboxymaltose (FCM) Cohort I | Iron Sucrose Cohort I | Ferric Carboxymaltose (FCM) Cohort II | Iron Dextran Cohort II
Number analyzed (Participants) | 10 | 8 | 10 | 9
mg
  Carbonyl | 11.69 (36.43) | -24.03 (65.55) | -18.20 (45.92) | -12.10 (54.85)
  8-isoprostane | 263.52 (896.57) | -417.89 (1030.83) | -29.35 (56.88) | -58.04 (159.58)

ADVERSE EVENTS:
Time Frame: 1 year and 10 months
Groups:
- Iron Sucrose or Iron Dextran: Intravenous iron
  Iron Sucrose / Iron Dextran: One 500 mg dose of IV iron sucrose administered over 4 hours (Cohort I), or a 750 mg dose of IV iron dextran administered as a 25 mg test dose over 5 minutes followed by a 725 mg dose over 3 hours if no adverse reaction to test dose is observed after 60 minutes (Cohort II)
Arm/Group | Ferric Carboxymaltose (FCM) | Iron Sucrose or Iron Dextran
Serious Adverse Events (participants affected / at risk) | 0/24 | 2/25
Other Adverse Events (participants affected / at risk) | 6/24 | 10/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ferric Carboxymaltose (FCM) (N=24) | Iron Sucrose or Iron Dextran (N=25)
Anaphylactic Reaction (Immune system disorders) | 0 (0) | 2 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ferric Carboxymaltose (FCM) (N=24) | Iron Sucrose or Iron Dextran (N=25)
Nausea (Gastrointestinal disorders) | 1 (1) | 2 (2)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
Injection site bruising (General disorders) | 1 (1) | 0 (0)
Anaphylactic reaction (Immune system disorders) | 0 (0) | 2 (2)
Hypersensitivity (Immune system disorders) | 2 (2) | 2 (2)
Hypophosphataemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days